CLINICAL TRIAL: NCT04862091
Title: A Randomized, Open-Label, Multi-Center, Parallel Controlled Study Comparing the Serum Testosterone Levels in Patients With Metastatic Castration-Resistant Prostate Cancer After Oral Administration of Abiraterone Acetate Tablets (I) or ZYTIGA®
Brief Title: Comparative Study of Abiraterone Acetate Tablets (I) or ZYTIGA® in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABTL-PD-01
Record Dates: First submitted 2021-04-25; First posted 2021-04-27 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Intervention Model Description: Abiraterone Acetate Tablets (I) compared with ZYTIGA®
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abiraterone Acetate Tablets (I) (Experimental)
  Interventions: Drug: Abiraterone Acetate Tablets (I)
- ZYTIGA®. (Active Comparator)
  Interventions: Drug: ZYTIGA®

INTERVENTIONS:
Drug: Abiraterone Acetate Tablets (I) — Abiraterone Acetate Tablets (I)
  Arms: Abiraterone Acetate Tablets (I)
Drug: ZYTIGA® — ZYTIGA®
  Arms: ZYTIGA®.

SUMMARY:
To evaluate whether the efficacy of the abiraterone acetate tablets (I) is comparable to that of the ZYTIGA®) by comparing the serum testosterone concentrations on Day 9 and/or Day 10 after oral administration of the two formulations in patients with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

1. Males, ≥ 18 years old;
2. Histologically or cytologically diagnosed with prostate adenocarcinoma, without neuroendocrine or small cell characteristics, and having metastatic lesions with imaging evidence (such as positive bone scan or metastatic lesions on CT/MRI);
3. Serum testosterone level < 50 ng/dL or 1.7 nmol/L at the screening; subjects who have not undergone bilateral orchidectomy must plan to continue medication throughout the study to maintain therapy with effective GnRH agonist or antagonist;
4. Progression of prostate cancer as confirmed by diagnostic files, meeting one of the conditions for disease progression: 1) Biochemistry evidence of recurrence: continuous 3 rises of PSA (taken a minimum of 1 week apart) from a baseline measurement of at least 2 ng/mL, greater than 50% of the minimum value in 2 rises; 2) Radiographic progression: a clear evidence of new lesion; 2 or more new bone lesions appearing on bone scan; CT or MRI showing lesion progression (RECIST 1.1);
5. ECOG performance status score of ≤ 1;
6. Life expectancy of ≥ 6 months;
7. Major organs are functioning well

Exclusion Criteria:

1. History of pituitary or adrenal dysfunction;
2. Have used flutamide within 4 weeks before the first dose of study treatment, and bicalutamide or nilutamide within 6 weeks before the first dose of study treatment;
3. Prior therapy with CYP17 inhibitors (such as abiraterone acetate, ketoconazole, TAK-700, etc.) or investigational drugs or marketed drugs of new androgen receptor antagonists (such as enzalutamide, apalutamide, SHR3680, ODM-201, and proxalutamide);
4. Have received 5-reductase inhibitors (such as finasteride and dutasteride), estrogen, progesterone, any herbal products (such as saw palmetto) that may decrease PSA levels, and radiotherapy within 4 weeks prior to the start of study medication;
5. Have previously received biotherapy or cytotoxic chemotherapy for mCRPC; patients who have completed docetaxel treatment for at least 1 year before enrollment can participate in screening;
6. Prostate cancer with moderate to severe pain symptoms, with a score of > 3 for Question 3 (the worst pain in the last 24 hours, 0-1 point means asymptomatic, 2-3 points mean mild symptoms) of the Brief Pain Inventory-Short Form (BPI-SF);
7. With contraindications to the use of glucocorticoids, such as uncontrolled persistent infections or other conditions;
8. Chronic diseases that require systemic corticosteroid therapy (> 10 mg/day prednisone or equivalent). Patients who have discontinued the administration or reduced the dose to < 10 mg within 14 days prior to the start of study treatment are eligible;
9. Presence of abdominal fistula, gastrointestinal perforation, abdominal abscess, or other abnormal gastrointestinal function within 6 months before the first dose of study treatment, which may affect drug absorption as judged by the investigator;
10. Presence of active heart disease within 6 months prior to the first dose of study treatment, including: severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, left ventricular ejection fraction < 50%, and severe arrhythmia requiring treatment or New York Heart Association (NYHA) Class III-IV heart failure;
11. Inability to swallow the whole tablet;
12. Other conditions that make the patient unsuitable for the study as judged by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Serum testosterone concentration | Day 9/Day 10
  Blood Sample tested for Serum Testosterone Levels

SECONDARY OUTCOMES:
PSA level | Day 28, Day 56, and Day 84
  The serum total PSA level
PSA-50 response rate | Day 28, Day 56, and Day 84
  The percentage of subjects with total serum PSA level decreased by 50% from the baseline value.
Absolute testosterone concentration | Day 9/10, Day 28, Day 56, and Day 84
  The actual measured serum testosterone concentration.
Testosterone inhibition rate | Day 9/10, Day 28, Day 56, and Day 84
  The percentage of subjects with a serum testosterone concentration of ≤ 1 ng/dL
Steady-state minimum concentration of abiraterone | Day 9/10, Day 28, Day 56, and Day 84
  Defined as the plasma concentration of abiraterone
Cmax, ss | Day 9
  Defined as the steady-state maximum concentration
AUC0-τ | Day 9
  Defined as the area under the curve within the dosing interval at steady state
Cmin, ss | Day 9
  Defined as the steady-state minimum concentration
Cav, ss | Day 9
  Defined as the mean blood drug concentration during the dosing interval at steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Lu X, Dai T, Chen X, Wu B, Chen H, Wu J, Yu D, Ge H, Li J, Huang H, Fan T, Cheng L, Zhang X, Zhang X, Yao X, Wei J, Xu Z, Yang W, He C, Luo J, Guan L, Fu B, Wang Q, Chen X, Zhang Y, Shi B, Zheng B, Wang Y, Luo H, Chen G, Wang H, Wang Q, Ye D. A randomized, open-label, multi-center, active-controlled phase II study comparing abiraterone acetate tablets (II), an improved formulation, versus originator abiraterone acetate in patients with metastatic castration-resistant prostate cancer. BMC Med. 2025 May 9;23(1):271. doi: 10.1186/s12916-025-04053-7. PMID 40346626